CLINICAL TRIAL: NCT04432389
Title: Phase IIb, Placebo-Controlled, Randomized, Double-Blind, Multicenter Study to Assess the Efficacy and Safety of Allogeneic Osteoblastic Cells (ALLOB®) Single Implantation in Tibial Fracture
Brief Title: Study to Assess the Efficacy and Safety of Allogeneic Osteoblastic Cells (ALLOB®) Single Implantation in Tibial Fracture
Acronym: ALLOB-TF2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bone Therapeutics S.A (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000013/BT
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALLOB (Experimental): Single injection of ALLOB at fracture site (4 ml)
  Interventions: Biological: ALLOB
- placebo (Placebo Comparator): Single injection of Placebo at fracture site (4 ml)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: ALLOB — After thawing, ALLOB® is a ready-to-use product for local administration at fracture site.
  Arms: ALLOB
Other: placebo — Placebo injected is a saline solution injectable grade (4 mL of 0.9% NaCl) filled in single-dose vial
  Arms: placebo

SUMMARY:
Although the majority of tibial fractures heal normally, some fractures may not heal within the usual time frame and is known as delayed bone healing within 4 to 6 months and absence of bone healing within 9 to 12 months in the most severe case of. Several factors can increase the risks of delayed healing complications like, for example, smoking, violent shocks (for example, due to a road accident) or even the type of fracture (an open fracture). The location of the fracture is also an important factor: among the bones of the arms and legs, the tibia is known for being the most at risk for complications. At tibial fracture with several risk factors could lead to delayed complications and interfere with patient daily life and reduce the quality of life.

The study drug, ALLOB®, is constituted of bone cells produced from the bone marrow of healthy adult donors. Preclinical studies have shown that ALLOB® cells are capable of forming bone and repairing fractures. When directly injected into a fracture, ALLOB® should therefore promote the healing of the fracture by re-establishing a healthy environment and stimulating bone production. To date, there is no treatment for fractures considered at risk of delayed complications. The current practice on diagnosis of complications is to wait at least 6-12 months before considering alternative interventions to promote fracture healing. The injection of ALLOB® quickly after the fracture should stimulate bone healing, reduce healing time, reduce complications, and improve the quality of life for the patient. ALLOB® has already shown preliminary evidence of effectiveness in the treatment of delayed bone healing fractures (ALLOB-DU1 clinical trial), including tibial fractures (8 patients). With this study, the Sponsor will evaluate whether ALLOB® promotes the healing of tibial fractures compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age
2. Subject diagnosed with a fresh proximal, midshaft or distal tibial fracture with definitive reduction performed with nail(s) and wound closure within 1 week of fracture occurrence
3. Mechanism of injury at risk of DU/NU: fracture occurring because of a high energy impact
4. At increased risk of DU/NU defined by:

   * Severe open fracture (Gustilo-Anderson grade IIIa and IIIb) OR
   * Open (Gustilo-Anderson grade I-II) or closed (Tscherne grade II-III) fracture with at least one additional risk factor among smoking , comminuted fracture or cortical continuity (0-50%)
5. Ability to obtain a written, dated, and signed informed consent prior to any study related procedures and ability to understand and comply with study requirements

Exclusion Criteria:

1. Definitive reduction at the fracture site under investigation performed with plate, screw or external fixator
2. Subjects who did not receive a standard antibiotic prophylaxis before definitive reduction at the fracture site under investigation
3. Intra-articular tibial pilon and/or plateau fracture at the site under investigation
4. Known osteomyelitis at the fracture site under investigation
5. Bone defect post-definitive reduction greater than 1cm at least on 2 cortices at the fracture site under investigation
6. Fracture requiring vascular surgery at the site under investigation
7. Pathological fractures as judged by the Investigator, such as tumor or metabolic bone disease
8. Bifocal or multifocal fracture at the site under investigation
9. Presence of fever (defined as body temperature ≥ 38°C) or other signs/symptoms suggestive of active infection before randomization
10. Severe brain trauma with a Glasgow Coma Scale (GCS) [3 - 8] or severe spinal cord injury with impossibility of weight-bearing
11. Current or history (within 5 years) of any neoplasia (except for basal cell carcinoma of the skin and for carcinoma in situ of the cervix that has been treated with no evidence of recurrence)
12. Known metabolic diseases potentially interfering with bone healing as judged by the Investigator, such as thyroid dysfunction, Paget disease or severe osteoporosis
13. Planned or history of solid organ transplantation or bone marrow transplantation
14. Known disease, including genetic disease, that may possibly need solid organ transplantation
15. Subject with renal impairment requiring dialysis or with clinically significant renal impairment defined as serum creatinine >2.0 x ULN
16. Clinically significant hepatic function impairment defined as ALT/AST levels > 3x ULN or total bilirubin levels > 2 x ULN
17. Known hematologic disease as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation
18. Subject with an history of long standing poorly controlled chronic hypertension or diabetes that could put him at risk of needing a kidney transplant later on according to the Investigator
19. History of hypersensitivity to human biological material including blood and blood derived products
20. Known allergy to DMSO, dextran, gentamicin and any other aminoglycosides
21. Participation in another interventional clinical study within 3 months prior to screening
22. Any chronic intake of medication within one month that might affect bone metabolism or the quality of bone formation such as but not limited to bisphosphonates, teriparatide, systemic steroids, anticoagulant therapies, methotrexate and other immunosuppressant drugs or related immunotherapy
23. Previous (within 10 years) treatment with bisphosphonates
24. Current treatment with bone morphogenic protein or any other osteo-biologic intervention at the site of the tibial fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects with a radiological success at Week 12 | 12 weeks
  A radiological success is defined as a subject with a Radiological Union Score for Tibia (RUST) above the threshold value predictive of a normal bone healing.

SECONDARY OUTCOMES:
Proportion of subjects with radiological success at Week 16, Week 20 and Month 6 | 16 weeks - 20 weeks - 6 months
  A radiological success is defined as a subject with a Radiological Union Score for Tibia (RUST) above the threshold value predictive of a normal bone healing.
Change in Radiographic Union Score for Tibia (RUST) at Week 12, Week 16, Week 20 and Month 6 compared to baseline visit | weeks 12 - 16 - 20 - 6 months
  Radiological fracture healing is defined by a radiological fracture union evaluated and adjudicated by Independent Radiologists.

CONTACTS AND LOCATIONS:
Locations (39):
- Belgium (4):
  - Tf2-Be-05, Anderlecht
  - Tf2-Be-03, Genk
  - Tf2-Be-04, Leuven
  - Tf2-Be-01, Lodelinsart
- Czechia (6):
  - Tf2-Cz-01, České Budějovice
  - Tf2-Cz-05, Jindřichův Hradec
  - Tf2-Cz-03, Kladno
  - Tf2-Cz-04, Nový Jičín
  - Tf2-Cz-02, Prague
  - Tf2-Cz-06, Prague
- France (5):
  - Tf2-Fr-06, Amiens
  - Tf2-Fr-04, Amiens
  - Tf2-Fr-01, Brest
  - Tf2-Fr-02, Chambray-lès-Tours
  - Tf2-Fr-06, Poitiers
- Germany (4):
  - Tf2-de-04, Giessen
  - Tf2-de-06, Lübeck
  - Tf2-de-02, Mannheim
  - Tf2-de-01, Münster
- Hungary (6):
  - Tf2-Hu-01, Budapest
  - Tf2-Hu-06, Eger
  - Tf2-Hu-05, Kaposvár
  - Tf2-Hu-02, Pécs
  - Tf2-Hu-03, Székesfehérvár
  - Tf2-Hu-04, Szolnok
- Poland (6):
  - Tf2-Pl-12, Kielce
  - Tf2-Pl-08, Krakow
  - Tf2-Pl-02, Lodz
  - Tf2-Pl-01, Szczecin
  - Ft2-Pl-07, Warsaw
  - Tf2-Pl-06, Warsaw
- Spain (8):
  - Tf2-Es-09, Badalona
  - Tf2-Es-08, Barcelona
  - Tf2-Es-02, Barcelona
  - Tf2-Es-03, Barcelona
  - Tf2-Es-07, Barcelona
  - Tf2-Es-06, Málaga
  - Tf2-Es-05, Pontevedra
  - Tf2-Es-01, Terrassa